CLINICAL TRIAL: NCT06234774
Title: Risk Factors for PPCs in Laparoscopic Non-Robotic vs Laparoscopic Robotic Abdominal Surgery (LapRas)- a Patient-Level Analysis of LAS VEGAS and AVATaR
Brief Title: Postoperative Pulmonary Complications in Robotic Versus Non-robotic Laparoscopic Surgery
Acronym: LapRas
Status: Completed | Type: Observational
Sponsor: University of Genova (Other)
Collaborators: University of Amsterdam (Other); University of Vienna (Other)
Responsible Party: Principal Investigator, Lorenzo Ball, Dr., University of Genova
Other Study IDs: LapRas
Record Dates: First submitted 2023-12-11; First posted 2024-01-31 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Respiratory Complication
Keywords: Postoperative pulmonary complications; Laparoscopic; Robotic Surgery; Mechanical Ventilation
MeSH Terms: interventions — Congresses as Topic; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robot-assisted surgery: Patients receiving abdominal surgical procedures with robot-assisted videolaparoscopic approach
  Interventions: Procedure: Robot-assisted laparoscopic surgery
- Non-robotic laparoscopic surgery: Patients receiving abdominal surgical procedures with conventional (non-robotic) videolaparoscopic approach
  Interventions: Procedure: Conventional (non-robotic) laparoscopic surgery

INTERVENTIONS:
Procedure: Robot-assisted laparoscopic surgery
  Groups: Robot-assisted surgery
Procedure: Conventional (non-robotic) laparoscopic surgery
  Groups: Non-robotic laparoscopic surgery

SUMMARY:
This secondary analysis aims to identify factors associated with the development of postoperative pulmonary complications (PPCs) in patients undergoing abdominal surgery, pooling and analyzing the data of two worldwide prospective studies, the 'Epidemiology, Practice of Ventilation and Outcome for Patients at Increased Risk of Postoperative Pulmonary Complications' (LAS VEGAS, NCT01601223) and the 'Assessment of Ventilatory management during general AnesThesia for Robotic surgery and its effects on postoperative pulmonary complications' (AVATaR, NCT02989415).

The primary aim is to compare the incidence of PPCs between patients undergoing non-robotic surgery versus patients undergoing robot-assisted surgery. One secondary aim is to determine which factors are associated with the occurrence of PPCs. The investigators hypothesize that differences in the occurrence of PPCs between the two surgery groups are more driven by differences in duration of anesthesia than by the intensity of ventilation.

DETAILED DESCRIPTION:
This study involves a preplanned analysis of a merged database comprising individual patient data from two global observational studies on ventilation and postoperative pulmonary complications (PPCs). Both study protocols, the LAS VEGAS and AVATaR were approved by a central Institutional Review Board and local ethics committees, with written informed consent obtained as per local legislation. The pooled database, including modifications for patient categories, does not require additional ethical approval or informed consent. The analysis will adhere to the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement.

Patients:

* The LAS VEGAS study includes patients undergoing general anesthesia with invasive ventilation for elective and non-elective surgeries.
* The AVATaR study includes patients aged over 18 undergoing robot-assisted surgery (RAS) for abdominal procedures.

Baseline Patient Characteristics:

- Key variables extracted from LAS VEGAS and AVATaR include demographic data, smoking status, comorbidities (chronic heart disease, obstructed sleep apnea syndrome, anemia, chronic kidney disease), and details about anesthesia and surgery.

Ventilation Variables:

* Ventilation-related variables extracted from the database include inspiratory pressure, plateau pressure, positive end-expiratory pressure, tidal volume, respiratory rate, fraction of inspired oxygen, peripheral oxygen saturation, end-tidal carbon dioxide.
* Mode of ventilation is classified as volume-controlled, pressure-controlled (including volume-guarantee pressure-controlled), and others.

Intensity of mechanical ventilation will be studied by three different estimators: the driving pressure, driving pressure multiplied by four plus respiratory rate and mechanical power.

For the statistical analysis medians with interquartile ranges, or as number with percentages, will be used as appropriate. Differences between the two groups of patients will be analyzes by Fisher or Wilcoxon test as appropriate. Key variables will be plotted by the cumulative distribution plots.

Numbers of available patients who meet inclusion criteria will represent our cohort of patients. The investigators estimated a 10 % of drop off for additional exclusion criteria. For this reason the enrollment of patients cannot be actual but just anticipated. The main analysis will be an univariable followed by a multivariable model including known risk factors for PPCs, intensity of ventilation and group (laparoscopic versus robotic surgery), covariates will be entered in the model. Logistic regression analysis will be performed for studying the association between PPCs and intensity of ventilation and duration of anesthesia. In case of relevant co-linearity of independent variables, separate models will be built excluding co-linear variables and the performances of the different models will be assessed using the corrected Akaike information criterion. In case of an association between RAS and PPCs: a mediation analysis to investigate the relationship between PPC and surgical approach will be conducted. In addition a matched-cohort analysis in patients with similar length of mechanical ventilation and intensity of ventilation will be performed. The mediation analysis will be reported according to the "A Guideline for Reporting Mediation Analyses" (AGReMA) statement. R Project for Statistical Computing will be used for analyzing data.

The analysis aims to compare incidences of PPCs after laparoscopic non-robotic and RAS abdominal surgeries, exploring associations with patient, surgery, and anesthesia factors.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients receiving invasive ventilation (via either an endotracheal tube or supraglottic device) during general anaesthesia for elective or non-elective surgery.

Exclusion Criteria:

* patients not undergoing laparoscopic surgery in LAS VEGAS, and not undergoing abdominal RAS in AVATaR;
* patients undergoing combined thoracic-laparoscopic surgery and patients in whom the intervention was converted from laparoscopic or RAS to open surgery are excluded;
* patients that received recent ventilation before surgery;
* patients with incomplete ventilation datasets not allowing the computation of intensity of ventilation, and patients with an incomplete follow-up for PPCs are also excluded.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients receiving invasive mechanical ventilation for laparoscopic or robot-assisted laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 2378 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | Postoperative day 5
  Composite end-point of post-operative pulmonary complications (new onset of acute respiratory distress syndrome (ARDS), pneumonia, pneumothorax, acute respiratory failure, need of oxygen therapy, need for postoperative invasive or non-invasive mechanical ventilation)

SECONDARY OUTCOMES:
Hospital length of stay | 1 year
  Days elapsed from surgery to discharge from hospital
In-hospital mortality | 1 year
  Death event occurring in the hospital after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Ball, MD PhD, Principal Investigator — University of Genova

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] LAS VEGAS investigators. Epidemiology, practice of ventilation and outcome for patients at increased risk of postoperative pulmonary complications: LAS VEGAS - an observational study in 29 countries. Eur J Anaesthesiol. 2017 Aug;34(8):492-507. doi: 10.1097/EJA.0000000000000646. PMID 28633157
- [Background] Assessment of Ventilation during general AnesThesia for Robotic surgery (AVATaR) Study Investigators; PROtective VEntilation (PROVE) Network; Writing Committee Members; Steering Committee Members; AVATaR Investigators. Ventilation and outcomes following robotic-assisted abdominal surgery: an international, multicentre observational study. Br J Anaesth. 2021 Feb;126(2):533-543. doi: 10.1016/j.bja.2020.08.058. Epub 2020 Oct 31. PMID 33131757